CLINICAL TRIAL: NCT00315432
Title: )A Study to Evaluate the Erythropoietic Response in HCV/HIV Co-Infected Patients Receiving Combination Ribavirin/Interferon Therapy
Brief Title: NATURAL HISTORY-Hepatitis C Virus/ Human Immunodeficiency Virus Coinfection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005134
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C; HIV; Anemia
Keywords: Natural History, Hepatitis C Infection, HIV Infection, HCV/HIV co-infection Ribavirin, Pegylated Interferon, Interferon
MeSH Terms: conditions — Hepatitis C; Anemia; HIV Infections | interventions — Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon and Ribavirin

SUMMARY:
The purpose of this study was to describe the time course and extent of hemoglobin (Hb) changes and the erythropoietic response to PEG-IFN/RBV (Pegylated Interferon and Ribavirin)-induced anemia In HCV(hepatitis C virus)/HIV (human immunodeficiency virus) co-Infected subjects.

DETAILED DESCRIPTION:
Patients receiving combination therapy for chronic hepatitis C virus (HCV) infection (standard or pegylated interferon alfa [PEG-IFN] in combination with ribavirin [RBV]) frequently develop moderate to severe anemia. In large, prospective, clinical trials of PEG-IFN alfa-2b and PEG-IFN alfa-2a, the reported mean decreases in hemoglobin (Hb) were 2.5 g/dL, and 3.7 g/dL, respectively. Furthermore, in a retrospective study, 54% of standard interferon/RBV-treated patients had hemoglobin decreases of at least 3 g/dL. It is important to understand the causes, natural history, and risk factors associated with HCV therapy-induced anemia, because such decreases in hemoglobin can result in RBV dose reduction or discontinuation, which may decrease the likelihood of a virologic response by patient. Erythropoietin is an endogenous hormone that acts in the bone marrow to increase the number of erythroid progenitor cells (red blood cells). Normally, a decrease in the hemoglobin level is accompanied by an increase in the serum erythropoietin (sEPO) level, which will ultimately normalize the Hemoglobin level. The relationship between hemoglobin and serum erythropoietin is less apparent in patients with chronic diseases such as cancer and human immunodeficiency virus (HIV) infection. It is not known whether HCV/HIV co-infected patients receiving combination PEG-IFN/RBV therapy have a similarly diminished erythropoietic response to anemia. The objective of this study is to document the pattern of hemoglobin changes and erythropoietic response (from baseline to final assessment) in HCV/HIV co-infected patients receiving combination therapy with IFN / RBV. N/A

ELIGIBILITY:
Inclusion Criteria:

* HIV- infected patients confirmed by HIV-RNA level
* HCV- infected patients confirmed by PCR(polymerase chain reaction) or branched DNA (b-DNA)
* Scheduled to commence combination IFN/RBV therapy on Day 1
* Normal serum creatinine
* On stable antiretroviral regimen (for HIV) for at least 4 weeks
* Life expectancy > 6 months

Exclusion Criteria:

* Patients with history of any primary hematologic disease
* Anemia attributable to factors such as iron or folate deficiency, pre-treatment
* hemolysis or gastrointestinal bleeding
* Has suspected or confirmed significant hepatic disease from an etiology other than
* HCV (e.g. alcohol, HBV DNA, autoimmune disease etc)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2000-09; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoints were change in hemoglobin and serum erythropoietin from baseline to week 8 (or early withdrawal)

SECONDARY OUTCOMES:
Other endpoints measured were changes in reticulocytes, platelets, total bilirubin, and RBV dose from baseline to week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Derived] Henry DH, Slim J, Lamarca A, Bowers P, Leitz G; HIV/HCV Coinfection Natural History Study Group. Natural history of anemia associated with interferon/ribavirin therapy for patients with HIV/HCV coinfection. AIDS Res Hum Retroviruses. 2007 Jan;23(1):1-9. doi: 10.1089/aid.2006.0082. PMID 17263626
- See also: A Study to Evaluate the Erythropoietic Response in HCV/HIV Co-Infected Patients Receiving Combination Ribavirin/Interferon Therapy or Ribavirin/PEG-Interferon — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=932&filename=CR005134_CSR.pdf